CLINICAL TRIAL: NCT04469920
Title: Evaluation of Pharmacokinetics and Safety of Saroglitazar Magnesium in Participants with Normal Hepatic Function and with Hepatic Impairment, Cholestatic Liver Disease, NASH with Advanced Fibrosis
Brief Title: Hepatic Impairment, Cholestatic Liver Disease, & NASH with Advanced Fibrosis & Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SARO.19.003
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — saroglitazar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1- mild hepatic impairment without evidence of PHT (Experimental): Subject with mild hepatic impairment without evidence of portal hypertension (PHT) based on Class A CPT score 5-6 points
  Interventions: Drug: Saroglitazar Magnesium 4 mg
- Group 2- mild hepatic impairment with evidence of PHT (Experimental): Subjects with mild hepatic impairment with evidence of portal hypertension based on Class A CPT score 5-6 points
  Interventions: Drug: Saroglitazar Magnesium 4 mg
- Group 3-moderate hepatic impairment (Experimental): Subjects with moderate hepatic impairment based on Class B CPT score 7-9 points
  Interventions: Drug: Saroglitazar Magnesium 4 mg
- Group 4- severe hepatic impairment (Experimental): Subjects with severe hepatic impairment based on Class C CPT score 10-14 points)
  Interventions: Drug: Saroglitazar Magnesium 4 mg
- Group 5-cholestatic liver disease (Experimental): Subjects with cholestatic liver disease
  Interventions: Drug: Saroglitazar Magnesium 2 mg; Drug: Saroglitazar Magnesium 4 mg
- Group 6-Non-cirrhotic Advanced Fibrosis secondary to NASH (Experimental): Subjects with Non-cirrhotic Advanced Fibrosis secondary to NASH
  Interventions: Drug: Saroglitazar Magnesium 2 mg; Drug: Saroglitazar Magnesium 4 mg
- Group 7- normal hepatic function (Experimental): Subjects with normal hepatic function
  Interventions: Drug: Saroglitazar Magnesium 2 mg; Drug: Saroglitazar Magnesium 4 mg

INTERVENTIONS:
Drug: Saroglitazar Magnesium 2 mg — 1 tablet, single dose at Day 1
  Other Names: Not any
  Arms: Group 5-cholestatic liver disease; Group 6-Non-cirrhotic Advanced Fibrosis secondary to NASH; Group 7- normal hepatic function
Drug: Saroglitazar Magnesium 4 mg — 1 tablet, single dose at Day 1
  Other Names: Not any

SUMMARY:
This will be a Phase 1, Open-label Study of Participants with Hepatic Impairment, Cholestatic Liver Disease, and NASH with Advanced Fibrosis and Normal Hepatic Function

DETAILED DESCRIPTION:
Male and female participants 18-80 years of age (inclusive) with normal hepatic function or hepatic impairment/disease who meet all of the inclusion and none of the exclusion criteria. Subjects with hepatic impairment will be enrolled based upon the Child-Pugh-Turcotte (CPT) classification system for mild hepatic impairment (Group 1 CPT Class A without PHT; Group 2 CPT Class A with PHT), moderate hepatic impairment (Group 3 Decompensated CPT Class B), or severe hepatic impairment (Group 4 Decompensated CPT Class C). Group 5 will include subjects with cholestatic liver disease and Group 6 will include subjects with non-cirrhotic advanced fibrosis secondary to NASH (non-alcoholic steatohepatitis). The control group (Group 7) will consist of demographic matched subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to comprehend and willingness to sign a written informed consent for the study.
2. Male or female aged 18 to 80 years (inclusive) at the time of signing the ICF.
3. Body mass index within the range 18.0 to 48.0 kg/m2 (inclusive) at screening.
4. Females must be non-pregnant, non-lactating and of non-childbearing potential or using highly efficient contraception for the full duration of the study.
5. Females of child-bearing potential and Males must agree to use contraception for the full duration of the study.
6. Ability to swallow and retain oral medication.
7. Groups 1 through 6 subjects may have medical findings consistent with their degree of hepatic dysfunction, as determined by medical history, physical examination, vital signs, ECGs, and clinical laboratory examinations at screening and check-in. Participants with abnormal findings considered not clinically significant by the Investigator are eligible.
8. Participants with hepatic impairment in Groups 1-4 will be classified at screening based on CPT score. If the hepatic impairment classification for the subject is not the same at screening and day -1, enrolment of the subject into a hepatic category group will be at the discretion of the hepatology Investigator.
9. Laboratory test values for Groups 1-4 hepatic impairment subjects must be clinically acceptable to the Investigator and meet all of the following parameters at Screening:

   1. ALT/AST value ≤ 10 × upper limit of normal (ULN)
   2. Absolute neutrophil count (ANC) ≥ 750/mm3
   3. Platelets ≥ 25,000/mm3
   4. Hemoglobin ≥ 8 g/dL
   5. α-fetoprotein < 50 ng/mL or 50-80 ng/mL with concurrent negative imaging study (US, CT, MRI)
10. Group 2 must have evidence of PHT as manifested by one of the following:

    1. presence of hepatic encephalopathy or ascites (on exam or imaging or medication to control these symptoms),
    2. historical or current presence of varices by imaging or endoscopy,
    3. historical or current presence of splenomegaly by imaging or physical exam,
    4. previous Hepatic Venous Pressure Gradient Measurement (HVPG) >10 mmHg,
    5. platelet count <150,000/mm3 (or /uL), or
    6. Fibroscan® at screening >20 kPa.
11. Documented history of cholestatic liver disease (i.e. primary biliary cholangitis, primary sclerosing cholangitis) OR alkaline phosphatase at screening of >1.25 x ULN with AST/ALT <1.2 x ULN OR Historical presence of AMA (anti-mitochondrial antibody) >1:40 and elevated alkaline phosphatase > ULN at screening
12. Clinical diagnosis of NASH and the following criteria:

    a. Screening Fibroscan® with liver stiffness > 8.5 kPa AND CAP >280 dB AND At least two criteria for metabolic syndrome modified from the NCEP

    ATP III Guidelines, at screening:

    i. Fasting glucose >100 mg/dL or receiving drug treatment for elevated glucose, ii. Fasting HDL cholesterol <40 mg/dL in men and <50 mg/dL in women or receiving drug treatment for low HDL cholesterol, iii. Fasting triglycerides > 150 mg/dL or receiving drug treatment for hypertriglyceridemia, iv. Waist circumference >102 cm for men or >88 cm for women or BMI >30 kg/m2, v. Systolic blood pressure >130 mmHg or diastolic blood pressure >85 mmHg or receiving drug treatment for hypertension

    OR:

    b. A historical liver biopsy within 6 months of screening consistent with NASH with stage 3 fibrosis and no documented weight loss >10% since date of liver biopsy
13. Subjects with normal hepatic function must match in age (± 10 years), gender, and weight (± 10 kg) with hepatic disease participants in the Groups 1-6.
14. Subjects should be in good health as determined by no clinically significant findings in the medical history, physical examination, vital signs, 12-lead electrocardiograms (ECGs), or laboratory examinations at Screening or Check-in.
15. Laboratory test values within normal limits or considered not clinically significant by the Investigator for subjects with normal hepatic function including ALT/AST < 1.2 × ULN at screening.

Exclusion Criteria:

1. Any significant, unstable medical condition or other instability that would prevent the subject from participating in the study as determined by the Investigator or designee.
2. History of malignancy of any type in the last 3 years of screening, with the exception of the following: in situ cervical or breast cancer or surgically excised non-melanoma skin cancers (i.e. basal cell or squamous cell carcinoma).
3. History of stomach or intestinal surgery or resection within the six months prior to screening that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, cholecystectomy, and hernia repair will be allowed).
4. History of any significant drug allergy (such as anaphylaxis) deemed clinically relevant by the Investigator.
5. Any major surgery within 3 months of screening.
6. Donation of blood or blood products within 3 months prior to screening.
7. Current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment or symptoms of active infectious disease within the two weeks prior to screening.
8. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, within 21 days prior to screening, unless deemed acceptable by the Investigator.
9. Receiving or has received any investigational drug within the 30 days or 5 halflives (whichever is longer), before receiving Saroglitazar Magnesium.
10. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2 by modification of diet in renal disease (MDRD) formula at screening.
11. Positive alcohol breath test at the time of check-in or those subjects who have current alcohol or substance abuse judged by the Investigator to potentially interfere with subject compliance or subject safety.
12. Positive test for drugs of abuse at screening or admission.
13. Any subject with poor peripheral venous access
14. Receipt of blood products within 1 month prior to check in.
15. Human immunodeficiency virus (HIV) type 1 antibody positive at screening for all groups.
16. Subjects who have had a change in hepatic disease status within 30 days of screening, as documented by the participant's medical history and deemed clinically significant by the Investigator.
17. Electrocardiogram QTcF > 500 msec, confirmed by repeat measurement OR presence of second- or third-degree atrioventricular (AV) block.
18. Subjects having -

    1. History of gastrointestinal bleeding within 1 month prior to screening.
    2. Current functioning organ transplant.
    3. Evidence of severe ascites requiring frequent paracentesis in the opinion of investigator.
19. Subjects having a history of any of the following: hepatic encephalopathy, ascites, history or current presence of varices by imaging or endoscopy, history or current presence of splenomegaly by imaging or physical exam, previous HVPG >10, platelet count <150,000 (or /uL) at screening, or Fibroscan® at screening >20 kPa.
20. QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 msec, confirmed by repeat measurement OR presence of second- or third-degree AV block.
21. Hepatitis B virus surface antigen (HBsAg) positive, Hepatitis C virus antibody (HCV-Ab) positive.
22. Subjects who use or intend to use any over the counter (vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) or prescription medications within 30 days or 5 half-lives (whichever is longer) prior to enrolment, with the exception of hormone replacement therapy and therapies for hepatic disease and treatments of associated disorders that have been stable for at least 30 days prior to screening and until Day 1, unless deemed acceptable by the Investigator (or designee).
23. Other known cause of liver disease such as NASH, Alcoholic Steatohepatitis (ASH), autoimmune hepatitis, or acute or chronic viral hepatitis as determined by the Investigator and subject's medical records
24. Evidence of liver decompensation such as ascites, hepatic encephalopathy or prior history of variceal bleed.
25. No other known cause of liver disease such as Primary Biliary Cholangitis (PBC), Primary Sclerosing Cholangitis (PSC), Alcoholic Steatohepatitis (ASH), autoimmune hepatitis, or acute or chronic viral hepatitis as determined by the Investigator and subject's medical records
26. Platelet count <150,000 (or /uL)
27. Subjects who have taken any prescription medications or over-the-counter medications, including herbal products, within 14 days prior to start of study drug dosing, with the exception of vitamins, acetaminophen, hormonal contraceptive medications and/or any other over-the-counter product approved by the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
AUC from time zero to infinity (AUC0-∞) | Before dosing on Day 1 through Day 7
  The area under the plasma concentration versus time curve from zero to infinity will be calculated by adding Ct/Kel to AUCt, where Ct is the last quantifiable concentration and Kel is the elimination rate constant.
AUC from time zero to the last quantifiable concentration (AUC0-t) | Before dosing on Day 1 through Day 7
  The area under the plasma concentration versus time curve will be calculated using the linear trapezoidal rule from the zero time point to the last quantifiable concentration.
Cmax | Before dosing on Day 1 through Day 7
  Maximum measured plasma concentration over the time span specified.
Tmax | Before dosing on Day 1 through Day 7
  Time of the maximum measured plasma concentration.
t1/2 | Before dosing on Day 1 through Day 7
  The half-life will be calculated by the equation tHalf = 0.693/ Kel. Kel (The terminal elimination rate constant) will be obtained from the slope of the line, fitted by linear least squares regression, through the terminal points of the natural log of the concentration versus time plot for these points
CL/F | Before dosing on Day 1 through Day 7
  Clearance
Vz/F | Before dosing on Day 1 through Day 7
  Volume of distribution

SECONDARY OUTCOMES:
Urine Pharmacokinetic: Ae | Before dosing on Day 1 through Day 5
  Amount of drug excreted during each collection interval
Incidence of AEs | Before dosing on Day 1 through Day 12
  Incidence and severity of AEs as a measure of safety and tolerability will be measured and reported.
Unbound Fraction | Day 1
  Unbound fraction in plasma of Saroglitazar
Unbound concentration | Day 1
  Unbound concentration in plasma of Saroglitazar

CONTACTS AND LOCATIONS:
Overall Officials: Deven Parmar, MD, Study Director — Zydus Therapeutics Inc.
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No